CLINICAL TRIAL: NCT01499589
Title: Can the Usage of Regional Block Room Save the Time of Anesthesia Team in the Main Orthopedic Operating Room?
Brief Title: Can the Usage of Regional Block Room Save the Time of Anesthesia Team
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Si562/2011
Record Dates: First submitted 2011-12-07; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Anesthesia; Time
Keywords: anesthesia-controlled time; turnover time
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- RA in block room: Performing regional anesthesia in the block room
  Interventions: Procedure: regional anesthesia
- RA inside OR: Performing regional anesthesia inside the main orthopedic operating room
  Interventions: Procedure: regional anesthesia

INTERVENTIONS:
Procedure: regional anesthesia — regional anesthesia procedure
  Other Names: neuraxial block; peripheral nerve block

SUMMARY:
Study of time usage of anesthesia team inside the main operating room compares between 2 groups of

* Performing regional anesthesia inside the operating room
* Performing regional anesthesia in the block room

Study purpose: How much will the investigators save time in the main operating room if we perform the regional anesthesia in the block room?

DETAILED DESCRIPTION:
Anesthesia-controlled time means anesthesia pre-procedure time plus anesthesia post-procedure time.

We also compares the anesthesia-controlled time in 3 groups of

* general anesthesia
* regional anesthesia
* general anesthesia combined with regional anesthesia

ELIGIBILITY:
Inclusion Criteria:

* elective orthopedic surgical patients that require for anesthesia ( start 9AM-4PM)

Exclusion Criteria:

* surgery under local infiltration

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: elective orthopedic surgical patients that require for anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
anesthesia-controlled time | 3 months
  anesthesia-controlled time = anesthesia pre-procedure time + anesthesia post-procedure time

SECONDARY OUTCOMES:
turnover time | 3 months
  turnover time = time new patient-in minus previous patient-out
number of elective cases after 4PM | 3 months
  number of the elective cases that will be running after 4 PM

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Tangwiwat, M.D, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand